CLINICAL TRIAL: NCT00320411
Title: Phase II Clinical Study of Lapatinib (GW572016) in Patients With ErbB2 Over - Expressing Advanced or Metastatic Breast Cancer
Brief Title: GW572016 In Patients With ErbB2 Over - Expressing Advanced Or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF104911
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Results first posted 2009-12-14 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms, Breast
Keywords: Stage IV breast cancer; Herceptin; metastatic breast cancer; ErbB1; ErbB2; trastuzumab; lapatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

ARMS (1):
- Lapatinb (Experimental): Lapatinib 1500mg QD
  Interventions: Drug: lapatinib

INTERVENTIONS:
Drug: lapatinib — Lapatinib 1500mg QD

SUMMARY:
This study (EGF104911) is designed to evaluate the efficacy and safety of lapatinib in patients with advanced or metastatic breast cancer. Eligible subjects must have ErbB2 overexpressing tumors and are refractory to treatment with anthracycline, taxanes and trastuzumab containing regimens. The study data obtained from EGF104911 will be combined with the data from EGF100642 and integrated analysis will be carried out in order to enhance the credibility of the study results.

ELIGIBILITY:
Inclusion Criteria:

A subject will be considered eligible for inclusion in this study only if all of the following criteria apply:

* Life expectancy of ≥16 weeks from the start of lapatinib therapy;
* Signed informed consent obtained from the patient;
* Subjects must have histologically confirmed breast cancer with advanced (Stage IIIb, IIIc with T4 lesion) or metastatic disease (including recurrent patients);
* Subjects must meet the following criteria regarding prior therapy:
* Anthracyclines, taxanes:
* If anthracycline- and taxane-containing regimens are administered sequentially;
* Subjects should have been provided with at least 2 cycles each and at least 4 cycles in total.
* If anthracycline- and taxane-containing regimen are administered concurrently;
* Subjects should have been provided with at least 4 cycles in total. or
* Subjects should have been provided with at least 2 cycles in total and provided progressive disease occurred.
* If anthracycline- and taxane-containing regimen are administered separately;
* Subjects should have been provided with at least 4 cycles each. or
* Subjects should have been provided with at least 2 cycles each and provided progressive disease occurred each regimen.
* Trastuzumab:
* Prior treatment must contain trastuzumab alone or in combination with other chemotherapy for at least 6 weeks of standard doses.
* Subjects must meet the following criteria regarding ErbB2 expression (defined by the following status before undergoing trastuzumab therapy.)

Patients with ErbB2 overexpression:

* 3+ by IHC, or FISH+
* 2+ by IHC and FISH+ are also eligible. However, patients with "2+ by IHC" who have previously been treated with trastuzumab should undergo FISH before study entry, if they have not had this test performed before, and are considered eligible only if their tumours are categorised as FISH+.
* Documentation of tumor progression or relapse after the most recent treatment is required.
* Archived tumor tissue must be available to compare tumor response with intra-tumoral expression levels of biomarkers (ErbB1 and ErbB2).
* Measurable lesion(s) according to RECIST (Response Evaluation Criteria in Solid Tumors); (See "6.3. Efficacy")
* A female, ≥20 and ≤74 years (at the time of giving consent), is eligible to enter and participate in this study if she is of:
* Non-childbearing potential (i.e., women with functioning ovaries who have a current documented tubal ligation or hysterectomy, or women who are post-menopausal, i.e., at least 1 year has past since the last menstrual period); or is
* The subject has a negative serum pregnancy test at screening, and agrees to one of the following from 2 weeks prior to administration of the first dose of lapatinib until 28 days after the final dose of lapatinib＊.
* Complete abstinence from intercourse:
* Consistent and correct use of one of the following acceptable methods of birth control:
* Injectable progestogen;
* Any intrauterine device (IUD);
* Oral contraceptives (either combined or Progestogen only);
* Barrier methods including diaphragm or condom with a spermicide.
* At least 3 weeks since the last dose of prior last chemotherapy, immunotherapy, biologic therapy, hormonal therapy, or radiotherapy (except for local radiation therapy to pain relief) for cancer or since the date of completion of surgery (except for minor surgical procedures) before beginning treatment with lapatinib, except for trastuzumab which must be discontinued at least 2 weeks prior to beginning of study drug. Subjects must have recovered or stabilized sufficiently from side effects associated with prior therapy;
* Prior to enrollment, radiation therapy is allowed to a limited field (e.g. painful bone mets, painful lumps), if it is not the sole site of measurable and/or assessable disease. Patients must have completed treatment and adequately recovered, in particular from bone marrow suppression.
* Subjects who are not on bisphosphonate therapy. Bisphosphonates initiated prior to study medication are allowed; however, initiation of bisphosphonate following the first dose of study medication is not allowed. Prophylactic use of bisphosphonates is only permitted for treatment of osteoporosis.
* Subjects with stable CNS metastasis (asymptomatic and off systemic steroids and anticonvulsants for at least 3 months) are also eligible;
* ECOG Performance Status of 0 to 2;
* Able to swallow and retain oral medication;
* Left ventricular ejection fraction (LVEF), measured by echocardiogram (ECHO), above the institutional's lower limit of normal (LVEF of ≥50% in such case as normal range of LVEF is not provided by institution).
* Subjects must have adequate organ function as defined below:
* Myelofunction:

Neutrophil count ≥1500 /mm3 Hemoglobin ≥9 g/dL (at least 2 weeks after blood transfusion if needed) Platelet count ≥100,000 /mm3

* Hepatic function:

Albumin ≤2.5 g/dL Total bilirubin ≤1.5xULN AST, ALT: ≤3xULN (without liver metastases), ≤5xULN (if documented liver metastases)

* Renal function:

Serum creatinine ≤1.5 mg/dL, or creatinine clearance ≤40 mL/min (calculated by the Cockcroft and Gault Method)

* Subjects who can visit the hospital once weekly (±3 days) at least in the first month after the start of lapatinib therapy and then every 4 weeks (±1 week) until the last assessment.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Pregnant or lactating females;
* Malabsorption Syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded;
* History of other malignancy. Subjects who have been disease free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible;
* Concurrent disease or condition that would make the subject inappropriate for study participation, or any serious medical disorder that would interfere with the subject's safety * [* ≥Grade 3 (according to NCI-CTCAE Version 3.0), as a general rule];
* Active or uncontrolled infection;
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure;
* Known history of or clinical evidence of leptomeningeal carcinomatosis;
* Participated in a clinical study within the past 28 days of the first dose of lapatinib;
* Prior therapy with an ErbB1inhibitor (e.g., gefinitib) and/or ErbB2 inhibitor other than trastuzumab;
* Has taken/received prohibited inhibitors (including foods) of CYP3A4 within 7 days prior to the first dose of study medication or has taken/received prohibited inducers inducers (including foods) of CYP3A4 within 14 days prior to the first dose of study medication(Refer to Appendix 7).
* The subject has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to lapatinib or excipients
* Patients ineligible for participation in the study in the judgment of the investigator/sub investigator.

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-11-28; Primary Completion 2009-04-01 (Actual); Study Completion 2009-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Japan (6):
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
- GSK Investigational Site

REFERENCES:
- [Background] Toi M, Iwata H, Fujiwara Y, Ito Y, Nakamura S, Tokuda Y, Taguchi T, Rai Y, Aogi K, Arai T, Watanabe J, Wakamatsu T, Katsura K, Ellis CE, Gagnon RC, Allen KE, Sasaki Y, Takashima S. Lapatinib monotherapy in patients with relapsed, advanced, or metastatic breast cancer: efficacy, safety, and biomarker results from Japanese patients phase II studies. Br J Cancer. 2009 Nov 17;101(10):1676-82. doi: 10.1038/sj.bjc.6605343. Epub 2009 Oct 20. PMID 19844234

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib Monotherapy: Lapatinib: 1500 mg (six 250 mg tablets) orally once daily
Period: Overall Study
Arm/Group | Lapatinib Monotherapy
Started | 62
Completed | 58
Not Completed | 4
Not completed — No investigational product admin. | 4

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 58

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumor Response
Description: Tumor response was measured as the number of participants achieving either a complete response (CR; disappearance of all target lesions) or partial response (PR; 30% decrease in the sum of the longest diameter of target lesions) among all participants who received study treatment. Tumor response was evaluated as the best response in accordance with response evaluation criteria in solid tumors (RECIST). Progressive disease: a 20% increase in the sum of the longest diameter of target lesions. Stable disease: small changes that do not meet the above-mentioned criteria.
Time Frame: Baseline and then followed every 4 weeks until disease progression or death. If treatment was terminated due to adverse events, then followed every 12 weeks until disease progression is noted.
Population: Intent-to-Treat (ITT) Population: all participants who had been registered and received at least one dose of the investigational product
Measure: Number; unit: participants
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 58
participants
  Complete response | 1
  Partial response | 8
  Stable disease | 18
  Progressive disease | 29
  Unknown | 2

2. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time between the point at which efficacy was noted until disease progression or death due to breast cancer.
Time Frame: First noted efficacy to disease progression; baseline and followed every 4 weeks until disease progression or death. If treatment was terminated due to adverse events, then followed every 12 weeks until disease progression is noted.
Population: Participants who achieved defined efficacy
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 9
weeks | 20.6 [16.1 to 32.1]

3. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time from the start of treatment until disease progression or death. Disease progression is defined as a 20% increase in the sum of the longest diameter of target lesions.
Time Frame: Baseline to disease progression or death; baseline and then followed every 4 weeks until disease progression or death. If treatment was terminated due to adverse events, then followed every 12 weeks until disease progression or death.
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 58
weeks | 8.4 [7.4 to 23.9]

4. Secondary Outcome: Clinical Benefit
Description: Clinical benefit was defined as the percentage of participants achieving complete response, partial response, and stable disease for more than 24 weeks.
Time Frame: Time at which all participants had been followed for at least 24 weeks; baseline and then followed every 4 weeks until disease progression (DP) or death. If treatment was terminated due to adverse events, then followed every 12 weeks until DP or death.
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 58
percentage of participants | 17.2
Statistical Analysis 1: Comparison: Lapatinib Monotherapy; Test type: Superiority or Other; percentage of participants = 17.2, 95% CI [8.6 to 29.4]

5. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from the start of treatment until first documented evidence of partial or complete tumor response (whichever status is recorded first).
Time Frame: Time at which all participants had been followed for at least 24 weeks; baseline and then followed every 4 weeks until disease progression (DP) or death. If treatment was terminated due to adverse event, then followed every 12 weeks until DP or death.
Population: Participants in the ITT Population achieving a partial or complete response
Measure: Median (Full Range); unit: Days
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 9
Days | 111 [56 to 279]

6. Secondary Outcome: 4-month Progression Free Survival
Description: The percentage of participants without progression or deaths at 4 months (16 weeks) after the start of dosing.
Time Frame: Baseline to Month 4 (Week 16)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 58
percentage of participants | 32.3
Statistical Analysis 1: Comparison: Lapatinib Monotherapy; Test type: Superiority or Other; percentage of participants = 32.3, 95% CI [20.0 to 44.7]

7. Secondary Outcome: 6-month Progression Free Survival
Description: The percentage of participants without progression or deaths at 6 months (24 weeks) after the start of dosing.
Time Frame: Baseline to Month 6 (Week 24)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 58
percentage of participants | 22.8
Statistical Analysis 1: Comparison: Lapatinib Monotherapy; Test type: Superiority or Other; percentage of participants = 22.8, 95% CI [11.6 to 34.0]

8. Secondary Outcome: Overall Survival
Description: Overall survival was measured as the time between the start of dosing until death, regardless of cause.
Time Frame: Start of dosing to death; baseline and then followed every 4 weeks until death while on treatment. If alive at time of treatment termination, then followed every 12 weeks until death.
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 58
weeks | 43.1 [24.3 to 80.7]

9. Secondary Outcome: Mean Phosphorylated 58 kDa Serine/Threonine Protein Kinase (p-AKT) H Score for All Participants
Description: Intra-tumoral expression levels of AKT, a tumor tissue biomarker, were measured using immunohistochemistry methods that incorporated both intensity and distribution of staining. A value designated the H score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+: 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum score of 0 to a maximum score of 300; the maximum score indicates the strongest expression.
Time Frame: Tumor samples taken at baseline
Population: Participants who provided enough tumor samples for this evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 10
units on a scale | 13.9 (26.32)

10. Secondary Outcome: Mean p-BAD H Score for All Participants
Description: Intra-tumoral expression levels of BAD, a tumor tissue biomarker, were measured using immunohistochemistry methods that incorporated both intensity and distribution of staining. A value designated the H score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+: 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum score of 0 to a maximum score of 300; the maximum score indicates the strongest expression.
Time Frame: Tumor samples taken at baseline
Population: Participants who provided enough tumor samples for this evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 9
units on a scale | 12.8 (36.50)

11. Secondary Outcome: Mean Bcl-2 H Score for All Participants
Description: Intra-tumoral expression levels of Bcl-2, a tumor tissue biomarker, were measured using immunohistochemistry methods that incorporated both intensity and distribution of staining. A value designated the H score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+: 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum score of 0 to a maximum score of 300; the maximum score indicates the strongest expression.
Time Frame: Tumor samples taken at baseline
Population: Participants who provided enough tumor samples for this evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 18
units on a scale | 20.9 (47.82)

12. Secondary Outcome: Mean Epidermal Growth Factor Receptor 3 (ErbB3) H Score for All Participants
Description: Intra-tumoral expression levels of ErbB3, a tumor tissue biomarker, were measured using immunohistochemistry methods that incorporated both intensity and distribution of staining. A value designated the H score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+: 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum score of 0 to a maximum score of 300; the maximum score indicates the strongest expression.
Time Frame: Tumor samples taken at baseline
Population: Participants who provided enough tumor samples for this evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 23
units on a scale | 185.5 (50.61)

13. Secondary Outcome: Mean Epidermal Growth Factor Receptor 4 (ErbB4) H Score for All Participants
Description: Intra-tumoral expression levels of ErbB4, a tumor tissue biomarker, were measured using immunohistochemistry methods that incorporated both intensity and distribution of staining. A value designated the H score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+: 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum score of 0 to a maximum score of 300; the maximum score indicates the strongest expression.
Time Frame: Tumor samples taken at baseline
Population: Participants who provided enough tumor samples for this evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 9
units on a scale | 133.3 (60.47)

14. Secondary Outcome: Mean Phosphorylated Extracellular Signal-regulated Kinase (p-ERK) H Score for All Participants
Description: Intra-tumoral expression levels of ERK, a tumor tissue biomarker, were measured.using immunohistochemistry methods that incorporated both intensity and distribution of staining. A value designated the H score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+: 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum score of 0 to a maximum score of 300; the maximum score indicates the strongest expression.
Time Frame: Tumor samples taken at baseline
Population: Participants who provided enough tumor samples for this evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 9
units on a scale | 12.2 (17.30)

15. Secondary Outcome: Mean Heregulin H Score for All Participants
Description: Intra-tumoral expression levels of Heregulin, a tumor tissue biomarker, were measured using immunohistochemistry methods that incorporated both intensity and distribution of staining. A value designated the H score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+: 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum score of 0 to a maximum score of 300; the maximum score indicates the strongest expression.
Time Frame: Tumor samples taken at baseline
Population: Participants who provided enough tumor samples for this evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 18
units on a scale | 55.3 (42.37)

16. Secondary Outcome: Mean Insulin-like Growth Factor 1 Receptor (IGF1R) H Score for All Participants
Description: Intra-tumoral expression levels of IGF1R, a tumor tissue biomarker, were measured using immunohistochemistry methods that incorporated both intensity and distribution of staining. A value designated the H score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+: 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum score of 0 to a maximum score of 300; the maximum score indicates the strongest expression.
Time Frame: Tumor samples taken at baseline
Population: Participants who provided enough tumor samples for this evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 23
units on a scale | 153.5 (48.44)

17. Secondary Outcome: Mean Survivin H Score for All Participants
Description: Intra-tumoral expression levels of Survivin, a tumor tissue biomarker, were measured using immunohistochemistry methods that incorporated both intensity and distribution of staining. A value designated the H score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+: 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum score of 0 to a maximum score of 300; the maximum score indicates the strongest expression.
Time Frame: Tumor samples taken at baseline
Population: Participants who provided enough tumor samples for this evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 10
units on a scale | 79.0 (47.25)

18. Secondary Outcome: Mean Terminal Deoxynucleotidyl Transferase Biotin-dUTP Nick End Labeling (TUNEL) H Score for All Participants
Description: Intra-tumoral expression levels of TUNEL, a tumor tissue biomarker, were measured using immunohistochemistry methods that incorporated both intensity and distribution of staining. A value designated the H score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+: 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum score of 0 to a maximum score of 300; the maximum score indicates the strongest expression.
Time Frame: Tumor samples taken at baseline
Population: Participants who provided enough tumor samples for this evaluation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lapatinib Monotherapy
Number analyzed (Participants) | 10
units on a scale | 48.9 (26.88)

ADVERSE EVENTS:
Arm/Group | Lapatinib Monotherapy
Serious Adverse Events (participants affected / at risk) | 14/58
Other Adverse Events (participants affected / at risk) | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Monotherapy (N=58)
Anorexia (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Pneumonia (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Hepatomegaly (Hepatobiliary disorders) | 1
Malaise (General disorders) | 1
Disease progression (General disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Ventricular dysfunction (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Monotherapy (N=58)
Diarrhea (Gastrointestinal disorders) | 36
Stomatitis (Gastrointestinal disorders) | 27
Nausea (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 2
Stomach discomfort (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 23
Pruritus (Skin and subcutaneous tissue disorders) | 13
Acne (Skin and subcutaneous tissue disorders) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 9
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Exfoliative rash (Skin and subcutaneous tissue disorders) | 5
Comedone (Skin and subcutaneous tissue disorders) | 5
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 4
Ingrowing nail (Skin and subcutaneous tissue disorders) | 4
Eczema (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin chapped (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Generalized erythema (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Asteatotic eczema (Skin and subcutaneous tissue disorders) | 1
Hair disorder (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Nasopharyngitis (Infections and infestations) | 13
Paronychia (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Eye lid infection (Infections and infestations) | 1
Localized infection (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Omphalitis (Infections and infestations) | 1
Fatigue (General disorders) | 23
Pyrexia (General disorders) | 11
Chest pain (General disorders) | 5
Malaise (General disorders) | 4
Edema (General disorders) | 3
Edema peripheral (General disorders) | 3
Pain (General disorders) | 3
Chest discomfort (General disorders) | 1
Ulcer (General disorders) | 1
Asthenia (General disorders) | 1
Weight decreased (Investigations) | 14
Alanine aminotransferase increased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 12
Blood alkaline phosphatase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 7
Hemoglobin decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 4
Blood urine present (Investigations) | 4
Blood uric acid increased (Investigations) | 2
White blood cell count decreased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 1
Eosinophil count decreased (Investigations) | 2
Neutrophil count increased (Investigations) | 2
White blood cell count increased (Investigations) | 2
Protein urine (Investigations) | 2
Blood urea increased (Investigations) | 2
Hematocrit decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Platelet count increased (Investigations) | 1
Blood albumin decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Blood glucose decreased (Investigations) | 1
Blood iron decreased (Investigations) | 1
Blood urea decreased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
Protein total decreased (Investigations) | 1
Weight increased (Investigations) | 1
Monocyte count increased (Investigations) | 1
Specific gravity urine (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 20
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 2
Hypoesthesia (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Hepatic encephalopathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 11
Mood altered (Psychiatric disorders) | 1
Anxiety disorder (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Cystitis-like symptom (Renal and urinary disorders) | 1
Abnormal sensation in eye (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eyelid edema (Eye disorders) | 1
Blepharospasm (Eye disorders) | 1
Scleral hemorrhage (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Conjunctival hyperemia (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Anemia (Blood and lymphatic system disorders) | 4
Lymph node pain (Blood and lymphatic system disorders) | 1
Iron deficiency anemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Flushing (Vascular disorders) | 4
Hot flush (Vascular disorders) | 2
Vasodilatation (Vascular disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Hepatic pain (Hepatobiliary disorders) | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 1
Nail avulsion (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Brachial plexus injury (Injury, poisoning and procedural complications) | 1
Seasonal allergy (Immune system disorders) | 2
Hypersensitivity (Injury, poisoning and procedural complications) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Genital hemorrhage (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Breast discharge (Reproductive system and breast disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Motion sickness (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.